CLINICAL TRIAL: NCT01588444
Title: Histological Comparison of Healing Following Tooth Extraction With Ridge Preservation Using Cortical Versus Cancellous Freeze Dried Bone Allograft
Brief Title: Ridge Preservation After Tooth Extraction Using Cortical Versus Cancellous Freeze Dried Bone Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20110039H
Record Dates: First submitted 2012-03-16; First posted 2012-05-01 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Tooth Extraction
Keywords: tooth extraction; bone grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cancellous FDBA (LifeNet) (Experimental): grafting with cancellous mineralized freeze-dried bone allograft (LifeNet Health)
  Interventions: Device: Cancellous FDBA
- cortical FDBA (LifeNet) (Experimental): CORTICAL FREEZE-DRIED BONE ALLOGRAFT (from LifeNet Health)
  Interventions: Device: cortical FDBA

INTERVENTIONS:
Device: cortical FDBA — cortical mineralized freeze-dried bone allograft
  Arms: cortical FDBA (LifeNet)
Device: Cancellous FDBA — CANCELLOUS FREEZE-DRIED BONE ALLOGRAFT (from LifeNet Health)
  Arms: cancellous FDBA (LifeNet)

SUMMARY:
The purpose of this study is to compare cortical and cancellous freeze-dried bone allograft (FDBA) materials in the preservation of alveolar bone following extraction of non-molar teeth. The primary objective is to histologically evaluate and compare the healing of extraction sockets of non-molar teeth grafted with cortical FDBA versus cancellous FDBA for ridge preservation.

ELIGIBILITY:
Inclusion Criteria:

* single rooted tooth requiring extraction with future dental implant placement

Exclusion Criteria:

* smoking > 10 cigarettes per day poorly controlled diabetes

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Mealey, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health Science Center Dental School, San Antonio, Texas, United States

REFERENCES:
- [Derived] Eskow AJ, Mealey BL. Evaluation of healing following tooth extraction with ridge preservation using cortical versus cancellous freeze-dried bone allograft. J Periodontol. 2014 Apr;85(4):514-24. doi: 10.1902/jop.2013.130178. Epub 2013 May 31. PMID 23725026

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cancellous FDBA (LifeNet) | Cortical FDBA (LifeNet)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patietns requring tooth extraction adn ridge preservation
Groups:
- Total: Total of all reporting groups
Arm/Group | Cancellous FDBA (LifeNet) | Cortical FDBA (LifeNet) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 53.4 [27 to 79] | 55.6 [31 to 69] | 54 [27 to 79]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Histologic Percentage of Vital Bone Formation
Description: Histologic percentage of vital bone formation in bone cores
Time Frame: 18-20 weeks after grafting
Measure: Median (Inter-Quartile Range); unit: percentage of vital bone
Arm/Group | Cancellous FDBA (LifeNet) | Cortical FDBA (LifeNet)
Number analyzed (Participants) | 20 | 20
percentage of vital bone | 12.98 [10.06 to 31.04] | 16.08 [12.12 to 30.25]

ADVERSE EVENTS:
Arm/Group | Cancellous FDBA (LifeNet) | Cortical FDBA (LifeNet)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes